CLINICAL TRIAL: NCT03922126
Title: Development of a Peer Intervention to Increase HIV/STI Testing and PrEP Uptake Among Latino Immigrant Men Who Have Sex With Men
Brief Title: Peer Intervention Latino Immigrant MSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Jane J. Lee, Assistant Professor, School of Social Work, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: STUDY00007054; KL2TR002317 (NIH)
Record Dates: First submitted 2019-04-15; First posted 2019-04-19 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: HIV Infections; Sexually Transmitted Diseases
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Listos peer intervention (Experimental): Listos intervention (peer counseling, PrEP information, and HIV/STI testing kits)
  Interventions: Other: Peer counseling; Diagnostic Test: HIV/STI self-testing kits
- Peer only group (Active Comparator): Peer only group (peer counseling, PrEP information)
  Interventions: Other: Peer counseling

INTERVENTIONS:
Other: Peer counseling — Information, motivation, and behavioral skills for HIV/STI testing and pre-exposure prophylaxis uptake
Diagnostic Test: HIV/STI self-testing kits — Kits to self-test for HIV/STIs
  Arms: Listos peer intervention

SUMMARY:
This study evaluates a peer intervention with HIV/STI self-testing kits to increase HIV/STI testing and PrEP uptake among Latino immigrant men who have sex with men. Half of participants will receive the "Listos" intervention (peer counseling, PrEP information, and HIV/STI testing kits) and half will receive the active control intervention (peer only group with no HIV/STI testing kits).

DETAILED DESCRIPTION:
HIV testing is crucial for early detection of HIV infection; yet, Latino immigrants are at high risk for late HIV diagnosis. Increased screening for HIV and STIs is particularly important for Latino immigrant men who have sex with men (MSM), a group disproportionately at risk for HIV that also encounters barriers to health access due to factors associated with immigrant status. Latino MSM recently experienced a significant increase (25%) in new HIV diagnoses (2008-2015), while diagnoses among MSM overall remained stable. Based on these trends, 1 in 4 Latino MSM will be diagnosed with HIV in their lifetimes, highlighting their urgent need for HIV prevention. Notably, pre-exposure prophylaxis (PrEP) can reduce risk of HIV among high-risk groups; yet, only 3% of Latinos who could benefit from PrEP have received it. As undiagnosed HIV contributes to 40% of new HIV infections, and STIs increase HIV risk, targeted interventions that address Latino immigrant MSM's barriers to HIV/STI testing and PrEP uptake are critical for curbing the HIV epidemic.

Studies have shown that peers can influence HIV-related behaviors by enhancing information, motivation, and behavior skills (IMB Model). Peers share characteristics with the target population, which facilitates role modeling and can empower individuals to engage in behaviors. While peer interventions have demonstrated success in shaping behaviors among Latino MSM, their utility for addressing immigrant-specific barriers to HIV/STI testing and PrEP use is less understood.

While the IMB Model and empowerment theory highlight relevant psychological determinants of behavior, competent attention to structural factors (i.e. access) is key for HIV prevention. The availability of HIV/STI self-testing kits presents opportunities to overcome structural barriers to testing. HIV/STI self-testing kits are convenient testing methods as they allow for at-home testing, reducing the need for health care visits. The research combines these approaches (peers and HIV/STI self-testing kits) to address individual and structural barriers to HIV prevention among Latino immigrant MSM.

ELIGIBILITY:
Inclusion Criteria:

* male sex (at birth)
* adult aged 18 and older
* immigrant (not born in continental U.S.)
* Latino (identifies as either Latinx or Hispanic
* reports sex with men in past 12 months
* reports not knowing their HIV status or being HIV negative

Exclusion Criteria:

* Does not identify as Latino/Hispanic
* Born in the continental U.S.
* Female sex (at birth)
* Does not report sex with men in the last 12 months
* Reports being HIV positive
* Younger than 18 years old

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Number of participants who test for HIV/STIs | 1 week
  Report of having tested for HIV or STIs
Number of participants who test for HIV/STIs | 6 weeks
  Report of having tested for HIV or STIs
Number of participants who test for HIV/STIs | 12 weeks
  Report of having tested for HIV or STIs
Number of participants who initiate PrEP | 1 week
  Report of use of PrEP
Number of participants who initiate PrEP | 6 weeks
  Report of use of PrEP
Number of participants who initiate PrEP | 12 weeks
  Report of use of PrEP

CONTACTS AND LOCATIONS:
Overall Officials: Jane J Lee, PhD, LMSW, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Lee JJ, Robles G, Leyva Vera CA, Orellana ER, Graham SM, Nguyen AM, Wei Y, Sanchez AH, Dombrowski JC, Simoni JM. A Peer-Based Intervention to Increase HIV and Sexually Transmitted Infection Testing Among Latinx Immigrant Sexual Minority Men in the US Pacific Northwest: Pilot Randomized Controlled Trial Conducted During the COVID-19 Pandemic. JMIR Form Res. 2023 Jul 12;7:e45871. doi: 10.2196/45871. PMID 37436792